CLINICAL TRIAL: NCT02608125
Title: A Phase I Open-Label, Multicenter, Dose-Escalation Study of PRN1371, a FGFR 1-4 Kinase Inhibitor, in Adult Patients With Advanced Solid Tumors, Followed by an Expansion Cohort in Patients With Metastatic Urothelial Carcinoma With FGFR 1, 2, 3, or 4 Genetic Alterations
Brief Title: A Dose Escalation Study in Solid Tumors and a Dose Expansion Study of PRN1371 in Adult Patients With Metastatic Urothelial Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: focus portfolio on immune-mediated diseases
Sponsor: Principia Biopharma, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRN1371-001
Record Dates: First submitted 2015-09-18; First posted 2015-11-18 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Solid Tumors; Metastatic Urothelial Carcinoma & Renal Pelvis & Ureter
Keywords: FGFR
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — PRN1371

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRN1371 (Experimental): Drug: PRN1371
  Interventions: Drug: PRN1371

INTERVENTIONS:
Drug: PRN1371

SUMMARY:
This is a multi-center, open label, non-randomized Phase 1 study, to be conducted in two parts, Part A, and Part B. Part A in solid tumors included the dose escalation phase for evaluating the safety and tolerability profile of PRN1371, a FGFR 1-4 Kinase inhibitor. Part B is the Cohort Expansion phase in patients with metastatic urothelial carcinoma to further evaluate safety and tolerability, preliminary activity, PK, and PD in patients with FGFR genetic alterations.

DETAILED DESCRIPTION:
The protocol specifies rules for dose-limiting toxicity and a maximum tolerated dose (MTD). To gain further experience with the MTD, and/or at some lower optimal biologic dose level, an expansion cohort (Part B) enrolled patients with metastatic urothelial carcinoma with fibroblast growth factor receptor (FGFR) 1, 2, 3 or 4 genetic alterations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological or cytological documentation of an advanced solid tumor
* Subject must have metastatic or recurrent disease and have failed first-line systemic treatment, and if indicated, failed approved second-line therapy, and for whom no standard therapy options are anticipated to result in a durable remission
* Subject must have evaluable, progressive, and measurable disease per the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines, Version 1.1
* Adequate bone marrow, liver, and renal function
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1

For Part B (expansion) in subjects metastatic urothelial carcinoma:

* The patient's tumor has been evaluated and prospectively identified as having FGFR 1, 2, 3, or 4 genetic alterations.

Exclusion Criteria:

* Patients who have received adequate prior treatment with a highly selective FGFR inhibitor
* Patients with other major uncontrolled medical conditions, e.g., recent myocardial infarction, stroke, diabetes, active hepatitis
* Patients who have received prior systemic anticancer therapy ≤ 3 weeks prior to study start (6 weeks for nitrosourea, antibodies, or mitomycin-C)
* Patients diagnosed with another primary malignancy within 3 years prior to study start, with the exception of adequately treated basal cell carcinoma, squamous cell carcinoma, or other non-melanomatous skin cancer, or carcinoma in situ of the uterine cervix
* Patients with glioblastoma multiforme
* Patient has a primary neoplasm of the brain or known uncontrolled metastases to the central nervous system (CNS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment related Grade 3 and/or Grade 4 adverse events, defined as dose limiting toxicities, for the doses of PRN1371 | 28 days on average

SECONDARY OUTCOMES:
Pharmacokinetic profile of PRN1371 including area under the serum concentration-time curve | Days 1 and 15
Pharmacokinetic profile of PRN1371 including maximum serum concentration | Days 1 and 15
Pharmacokinetic profile of PRN1371 including time to maximum serum concentration | Days 1 and 15
Pharmacodynamic profile of PRN1371 including the effect of PRN1371 on phosphate levels | While being treated with PRN1371 (expected average of 16 weeks)
Pharmacodynamic profile of PRN1371 including the effect of PRN1371 on calcium levels | While being treated with PRN1371 (expected average of 16 weeks)
Pharmacodynamic profile of PRN1371 including the effect of PRN1371 on serum FGF23 (Part A only) levels | While being treated with PRN1371 (expected average of 16 weeks)
Objective response rate (ORR) as measured by RECIST v1.1 in patients treated with PRN1371 | Every 8 weeks while being treated with PRN1371 (expected average of 16 weeks)
Duration of response in patients treated with PRN1371 | Every 8 weeks while being treated with PRN1371 (expected average 16 weeks)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - UCSF Helen Diller Family Comprehensive Cancer Cener, San Francisco, California
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Wake Forest University Health Sciences Medical Center, Winston-Salem, North Carolina
  - Tennessee Oncology, Sarah Canon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Spain (7):
  - Vall d'Hebron Institute of Oncology (VHIO), Vall d'Hebron University Hospital, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario Ramon y Cajal, Madrid
  - START Madrid-FJD Fundacion Jiminez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - START Madrid-CIOCC, Centro Integral Oncológico Clara Campal, Madrid
  - Hospital Virgen del Rocio, Seville